CLINICAL TRIAL: NCT06942585
Title: Acute Effects of Dynamic and Kinesiology Taping on Balance and Kinesthesia of the Lower Limbs in Healthy Adults
Brief Title: Effects of Dynamic and Kinesiology Taping on Balance and Kinesthesia in Healthy Adults
Acronym: DAKTIK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Primorska (Other)
Responsible Party: Principal Investigator, Žiga Kozinc, Assistant professor, University of Primorska
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: DAKTIK
Record Dates: First submitted 2025-04-08; First posted 2025-04-24 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Dynamic Tape; Kinesiology Taping

STUDY DESIGN:
Intervention Model Description: This study uses a randomized crossover design, where each participant serves as their own control. All participants will undergo three separate testing sessions in randomized order: (1) no tape, (2) kinesiology tape (KT), and (3) dynamic tape (DT). A washout period will be ensured between sessions to minimize potential carryover effects. This design allows for direct within-subject comparisons of the acute effects of KT and DT on balance and kinesthesia.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Kinesiology tape (Experimental): Kinesiology tape (KT) applied to the knee and ankle
  Interventions: Device: Kinesiology Tape
- Dynamic tape (Experimental): Dynamic tape (DT) applied to the knee and ankle
  Interventions: Device: Dynamic tape

INTERVENTIONS:
Device: Kinesiology Tape — An elastic therapeutic tape applied to the ankle and knee using standard kinesiology taping techniques. The tape is stretched to approximately 10-15% during application and is designed to mimic the properties of human skin. It aims to provide sensory stimulation, improve proprioceptive feedback, and support joint function without limiting range of motion. The application targets muscles and tendons surrounding the knee and ankle, commonly used in both preventive and rehabilitative physiotherapy.
  Arms: Kinesiology tape
Device: Dynamic tape — A biomechanical tape characterized by high elasticity (over 200%) and strong resistance, applied to the ankle and knee to assist movement and absorb load. The tape is applied in a shortened muscle position with maximal stretch across the joint, following the manufacturer's guidelines (GripIt ACTIVETAPE, 5 cm width). This taping method aims to provide both mechanical support and neurosensory input, facilitating muscle activation and improving joint stability during movement. It is used to address both biomechanical and proprioceptive components of lower limb control.
  Arms: Dynamic tape

SUMMARY:
This study aims to investigate the acute effects of dynamic tape (DT) and kinesiology tape (KT) on balance and kinesthesia of the lower limbs in healthy young adults. Participants will undergo assessments of static balance and knee joint position sense before and after the application of each taping condition. The study seeks to determine whether DT or KT can provide immediate improvements in postural stability and proprioceptive accuracy.

DETAILED DESCRIPTION:
Taping techniques are commonly used in rehabilitation and sports settings to support joint function, reduce pain, and improve proprioception. Dynamic tape (DT) and kinesiology tape (KT) differ in their mechanical properties and proposed mechanisms of action. While KT is elastic and mimics the properties of skin, DT offers higher elasticity and resistance, potentially providing enhanced mechanical support and proprioceptive feedback.

Although several studies have explored the effects of taping on balance and proprioception, direct comparisons between DT and KT, particularly when applied to both the ankle and knee joints, remain limited. This study seeks to address this gap by examining and comparing the immediate effects of DT and KT on static balance and kinesthesia of the lower limbs in healthy adults.

The findings may contribute to a better understanding of the clinical relevance of different taping methods and inform decision-making in preventive and therapeutic interventions targeting lower limb stability and proprioception.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18-30 years
* No current pain or injury affecting the lower limbs
* Willingness to participate and provide informed consent
* No known allergy or sensitivity to adhesive materials

Exclusion Criteria:

* History of ankle sprain or anterior cruciate ligament (ACL) injury
* Any lower limb injury in the past 3 months
* Neurological or vestibular disorders affecting balance
* Skin conditions or wounds at the taping sites
* Participation in balance or proprioception training programs in the past month

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-05-16 (Actual); Study Completion 2025-05-19 (Actual)

PRIMARY OUTCOMES:
Mean Velocity of Center of Pressure During Single-Leg Stance [mm/s] | Immediately before and within 10 minutes after tape application (per condition)
  Mean velocity of the CoP will be measured during the 30-second single-leg stance using a force plate. The outcome will be compared across the no tape, kinesiology tape, and dynamic tape conditions.
Sway Amplitude of Center of Pressure During Single-Leg Stance [mm] | Immediately before and within 10 minutes after tape application (per condition)
  During the same 30-second single-leg stance test, the sway amplitude of the CoP will be recorded using a force plate. This outcome will be used to evaluate changes in postural control across taping conditions.

SECONDARY OUTCOMES:
Knee Joint Kinesthesia [°] | Immediately before and within 10 minutes after tape application (per condition)
  Kinesthesia will be assessed using a passive-to-active joint position reproduction test with a digital goniometer (EasyAngle). Participants will attempt to replicate a reference knee flexion angle (45°) with eyes closed. The absolute angular error (in degrees) between the target and reproduced position will be calculated. Measurements will be compared across the no tape, kinesiology tape, and dynamic tape conditions to evaluate the acute effects of taping on proprioceptive accuracy.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Primorska, Faculty of Health Sciences, Izola, Izola, Izola, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) will not be shared due to the small sample size, the nature of the data (short-term, non-clinical outcomes), and to protect participant confidentiality. Aggregated results will be published in scientific outlets and shared upon request.